CLINICAL TRIAL: NCT06476756
Title: Combined Effects of Active Cycle Breathing Technique and Buteyko Technique on Airway Clearance in Post Sternotomy Patients
Brief Title: Combined Effects of Active Cycle Breathing Technique and Buteyko Technique in Post Sternotomy Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR & AHS/23/0375
Record Dates: First submitted 2024-06-12; First posted 2024-06-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Sternotomy
Keywords: Buteyko

STUDY DESIGN:
Intervention Model Description: Group A: combine effects of ACBT and Buteyko techniques will be performed first 3days of cardiac rehab phase 1.
  Group B: effect of buteyko techniques will be performed first three days of cardiac rehab phase 1.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACTIVE CYCLE OF BREATHING TECHNIQUE (Experimental): Group A: combine effects of ACBT and Buteyko techniques will be performed first 3days of cardiac rehab phase 1.
  Interventions: Other: ACTIVE CYCLE OF BREATHING TECHNIQUE
- Buteyko techniques (Experimental): Group B: effect of buteyko techniques will be performed first three days of cardiac rehab phase 1.
  Interventions: Other: Buteyko techniques

INTERVENTIONS:
Other: ACTIVE CYCLE OF BREATHING TECHNIQUE — Group A: combine effects of ACBT and Buteyko techniques will be performed first 3days of cardiac rehab phase 1.
  Arms: ACTIVE CYCLE OF BREATHING TECHNIQUE
Other: Buteyko techniques — Group B: effect of buteyko techniques will be performed first three days of cardiac rehab phase 1.
  Arms: Buteyko techniques

SUMMARY:
This randomized clinical trial seeks to compare the efficacy of the Active Cycle of Breathing Technique (ACBT) and Buteyko breathing techniques in sternotomy patients undergoing coronary artery bypass graft (CABG) surgery, aged 30 to 60. Data will be collected from Surgical Intensive Care Unit (ICU) in selected hospitals. Participants will be assigned to intervention to receiving ACBT and Buteyko breathing techniques standard protocol including chest percussion , tissue blowing exercises, incentive spirometer , cough technique, breathing control, deep breathing, and deep breathing techniques.

DETAILED DESCRIPTION:
This randomized clinical trial seeks to compare the efficacy of the Active Cycle of Breathing Technique (ACBT) and Buteyko breathing techniques in sternotomy patients undergoing coronary artery bypass graft (CABG) surgery, aged 30 to 60. Data will be collected from Surgical Intensive Care Unit (ICU) in selected hospitals. Participants will be assigned to intervention to receiving ACBT and Buteyko breathing techniques standard protocol including chest percussion , tissue blowing exercises, incentive spirometer , cough technique, breathing control, deep breathing, and deep breathing techniques. The three-day trial, starting upon ICU/CCU admission, will measure primary and secondary outcomes before and after each session for both groups. Statistical analysis using SPSS version 25 will be employed post data collection.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-60 years
* Patient underwent cardiac surgery for first time
* Having speaking, hearing, cognitive ability
* Both genders ( Male and female)
* On mechanical ventilation for less than 24h after surgery

Exclusion Criteria:

* • Hemodynamic ally unstable patients

  * Patients with reopening of sternum
  * Infection patients
  * Renal failure
  * Arrhythmia
  * Patient on mechanical ventilator
  * Cancer
  * Tuberculosis

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-03-10 (Actual); Primary Completion 2024-07-15 (Estimated); Study Completion 2024-08-20 (Estimated)

PRIMARY OUTCOMES:
Borg dyspnea scale | base line and 4 week
  The Borg RPE scale rates exertion from a scale of 6 (no exertion) to 20 (maximum effort). A rating between 12 to 14 typically reflects a moderate or somewhat hard level of intensity.
BREATHLESSNESS, COUGH AND SPUTUM SCALE (BCSS) | 4 weeks
  The BCSS is a three-item patient-reported questionnaire that rates sputum, cough, and dyspnea . This instrument can identify a disease aggravation with sensitivity and specificity.

CONTACTS AND LOCATIONS:
Overall Officials: Sidra Faisal, PP-DPT, Principal Investigator — Riphah International University
Locations (1):
- Gulab Devi teaching hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cappello IA, Candelari M, Pannone L, Monaco C, Bori E, Talevi G, Ramak R, La Meir M, Gharaviri A, Chierchia GB, Innocenti B, de Asmundis C. 3D Printed Surgical Guide for Coronary Artery Bypass Graft: Workflow from Computed Tomography to Prototype. Bioengineering (Basel). 2022 Apr 19;9(5):179. doi: 10.3390/bioengineering9050179. PMID 35621457
- [Background] Frak W, Wojtasinska A, Lisinska W, Mlynarska E, Franczyk B, Rysz J. Pathophysiology of Cardiovascular Diseases: New Insights into Molecular Mechanisms of Atherosclerosis, Arterial Hypertension, and Coronary Artery Disease. Biomedicines. 2022 Aug 10;10(8):1938. doi: 10.3390/biomedicines10081938. PMID 36009488
- [Background] Kamiya K, Takei M, Nagai T, Miyoshi T, Ito H, Fukumoto Y, Obara H, Kakuma T, Sakuma I, Daida H, Iimuro S, Shimokawa H, Kimura T, Nagai R, Anzai T. Association between Non-Lipid Residual Risk Factors and Cardiovascular Events in Patients with Stable Coronary Artery Disease Treated with Pitavastatin: An Observation from the REAL-CAD Study. J Atheroscler Thromb. 2024 Jan 1;31(1):61-80. doi: 10.5551/jat.64304. Epub 2023 Aug 11. PMID 37574272